CLINICAL TRIAL: NCT06184880
Title: Effect of Physical Activity Program on Sedentary and Physical Activity Level of Patients With Upper Aerodigestive Tract Cancer
Brief Title: Effect of Physical Activity Program on Sedentary of Patients With Upper Aerodigestive Tract Cancer
Acronym: APAORL2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valence (Other)
Collaborators: Claude Bernard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH-CHV-14
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Upper Aerodigestive Tract Cancer; Head and Neck Cancer
Keywords: Physical Activity; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: a randomized, open label, controlled, monocentric, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A control group (Active Comparator): Patients will receive standard care, recommendations on physical activity.
  patients should wear the wristband continuously for 7 days prior to scheduled hospital visit T0, T1, T2, T3, T4, T5
  Interventions: Behavioral: behavioral; Other: Sedentary
- B experimental Group (Experimental): 1 or 2 physical activity sessions per week, either face-to-face or by videoconference at patient convenience: low-to-moderate intensity aerobic and anaerobic muscle-strengthening session and a 40-minute stretching/yoga session.
  patients should wear the wristband continuously for 7 days prior to scheduled hospital visit T0, T1, T2, T3, T4, T5
  Interventions: Behavioral: behavioral; Other: Sedentary

INTERVENTIONS:
Behavioral: behavioral — International Physical Activity (IPAQ) Questionnaire, Quality of Life Questionnaire QLQ-C30, HN 43 questionnaire, Multidimensional Fatigue Inventory (MFI) Questionnaire, Big Five Inventory Questionnaire, illness Identity Questionnaire,
Other: Sedentary — Actimetry (cumulative time without movement over 24h, prolonged sedentary periods >30 min without movement. Continuous recording 7 days prior to visit T0, T1, T2, T3, T4, T5
  Other Names: Physical Activity level

SUMMARY:
APAORL2 study aims to evaluate the efficacy of a physical activity program on the sedentary and physical activity level during the 18-month program.

APAORL2 study is a randomized, open label, controlled, monocentric, intervention study that will be conducted among 96 patients treated for localized upper aerodigestive tract cancer.

DETAILED DESCRIPTION:
Rationale:

A sedentary lifestyle has been clearly shown to reduce survival in cancer patients, mainly through metabolic changes. While the notions of sedentary lifestyle and physical inactivity overlap, they are not entirely synonymous.

The aim of this study is to examine the contribution of a physical activity program, during the treatment and post-treatment phases, in addition to the current care program, on behavior change (i.e. sedentary behaviors and Physical activity levels), quality of life and fatigue in patients with upper aerodigestive tract cancer

The primary objective is to show that the experimental group (combining the current care pathway + physical Activity program) has lower levels of sedentary behaviour and higher levels of physical activity than the control group (following the classic care pathway with Physical Activity awareness) after the treatment phase.

Patients will be randomly assigned to one of the 2 arms of the study according to a 1:1 ratio:

Group A: control group: standard care with recommendations on physical activity.

Group B: experimental group: Physical activity program

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* newly diagnosed, histologically proven Upper Aerodigestive Tract Cancer, non-metastatic,
* life expectancy ≥18 months
* having a smartphone, tablet or computer with an internet connection enabling remote physical Activity sessions for the experimental group

Exclusion Criteria:

* Presenting a contraindication to moderate physical activity
* Deprived of their liberty by court or administrative decision
* Unable to be followed for medical, social, family, geographic or psychological reasons for the duration of the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
sedentary level | Change between baseline and 3, 6, 12 months and 18 months
  cumulative time without movement over a day, as well as prolonged sedentary periods (>30min without movement): continuous recording 7 days prior to hospital visits

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Change between baseline and 3, 6, 12 months and 18 months
  Physical Activity level
Quality of Life Questionnaire QLQ-C30 | Change between baseline and 3, 6, 12 months and 18 months
  Quality of Life
Head Neck (HN) 43 questionnaire | Change between baseline and 3, 6, 12 months and 18 months
  Quality of Life
Multidimensional Fatigue Inventory: MFI questionnaire | Change between baseline and 3 months
  fatigue level
Big Five Inventory questionnaire | Change between baseline and 3 months
  measure personality traits.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Guillaume, Principal Investigator — CH VALENCE

IPD SHARING:
Plan to Share IPD: No